CLINICAL TRIAL: NCT01294527
Title: Multicenter, Prospective Evaluation of Performance, Safety, and Surveillance of the WiCS-LV System in Patients Indicated for Cardiac Resynchronization Therapy
Brief Title: Wireless Stimulation Endocardially for Cardiac Resynchronization Therapy
Acronym: WiSE-CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EBR Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EBR-00980
Record Dates: First submitted 2011-02-08; First posted 2011-02-11 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Heart Failure; Ventricular Dysfunction; Cardiomyopathy
Keywords: Cardiac Resynchronization Therapy; cardiac pacing; electrical stimulation; bi-ventricular pacing
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction; Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Implant (Experimental): Implant of the WiCS-LV system
  Interventions: Device: Wireless cardiac stimulator implant to pace the left ventricle for CRT

INTERVENTIONS:
Device: Wireless cardiac stimulator implant to pace the left ventricle for CRT — Transvascular endocardial implantation of wireless pacing Electrode and subcutaneous implantation of Implantable Pulse Generator
  Other Names: WiCS-LV system

SUMMARY:
The WiCS-LV system is an alternative means to providing left ventricular stimulation for Cardiac Resynchronization Therapy (CRT). The purpose of this study is to evaluate the safety and performance of the WiCS-LV System in patients with indications for CRT.

DETAILED DESCRIPTION:
Eligible patients will undergo an acoustic window assessment using transthoracic echocardiography. Patients with adequate acoustic windows will undergo implantation of the WiCS-LV system.

Patients will undergo evaluations pre-hospital discharge, and at one month, 3 months, and 6 months post implantation. Extended follow-up will be obtained via a registry at 1, 2, 3, 4, and 5 years post implantation.

ELIGIBILITY:
Inclusion Criteria:

Patients with standard indication for CRT based upon the most recent guidelines AND meeting criteria for one of these three categories:

1. Patients with previously implanted pacemakers or ICD's and meeting standard indications for CRT - referred to as "upgrades"
2. Patients in whom attempted coronary sinus lead implantation for CRT has failed - referred to as "untreated"
3. Patients with previously implanted CRT device, not responding to CRT (no change or worsening of symptom or NYHA functional class after 6 months of treatment confirmed by investigator) - referred to as "non-responders"

Exclusion Criteria:

1. Inability to comply with the study follow-up or other study requirements
2. Contraindication to heparin
3. Contraindication to both chronic anticoagulants and antiplatelet agents
4. Contraindication to iodinated contrast agents
5. Intracardiac thrombus by transesophageal echocardiography
6. Age less than 18 years
7. Attempted IPG implant within 3 days
8. Life expectancy of < 12 months
9. Chronic hemodialysis
10. Myocardial infarction within one month
11. Major cardiac surgery within one month
12. Female of childbearing potential, pregnant, or breastfeeding
13. Noncardiac implanted electrical stimulation therapy devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-02; Primary Completion 2012-04 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with device-related adverse events as a measure of safety | 24 hour peri-operative and one month
  Device-related adverse events are those in which the WiCS-LV system is directly or indirectly responsible.
Number of patients with procedure-related adverse events as a measure of safety | 24 hour perioperative and one month
  Procedure-related adverse events are those which occur during the WiCS-LV system implant procedure.
Bi-ventricular pacing capture | one month
  Bi-ventricular pacing capture documented on 12-lead EKG

SECONDARY OUTCOMES:
Number of patients with device-related adverse events as a measure of safety | 6 months
  Device-related adverse events are those in which the WiCS-LV system is directly or indirectly responsible.
Number of patients with serious adverse events as a measure of safety | 6 months
Left ventricular pacing capture | 1, 3, and 6 months
  Left ventricular pacing capture documented on 12-lead EKG
Bi-ventricular pacing capture | 3 and 6 months
  Bi-ventricular pacing capture documented on 12-lead EKG
Bi-ventricular pacing capture | 1, 3, and 6 months
  Bi-ventricular pacing capture on 24 hour ambulatory monitoring
Clinical composite score | 6 months
  Composite of all cause mortality, heart failure hospitalization, NYHA class, and patient global assessment
Change in echocardiographic indices | 6 months
  change in left-ventricular end-systolic volume, left ventricular end-diastolic volume, and ejection fraction
Change in blood laboratory Brain Natriuretic Peptide | 6 months
  change in NT-proBNP level

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Auricchio, MD, Principal Investigator — Fondazione Cardiocentro, Lugano CH
Locations (10):
- France (2):
  - Nouvelles Clinicques Nantaises, Nantes
  - Hospital Pontchaillou-CHU, Rennes
- Germany (5):
  - Kerckhoff-Klinik, Bad Nauheim
  - Herzzentrum Brandenburg, Bernau
  - Klinium Coburg gGmbH, Coburg
  - Facharztzentrum Dresden-Neustadt GbR, Dresden
  - Herzzentrum Leipzig GmbH, Leipzig
- Netherlands (2):
  - Leiden University Medical Centre, Leiden
  - Isala Klinieken Zwolle, Zwolle
- Cardiocentro Ticini, Lugano, Switzerland

REFERENCES:
- [Derived] Auricchio A, Delnoy PP, Butter C, Brachmann J, Van Erven L, Spitzer S, Moccetti T, Seifert M, Markou T, Laszo K, Regoli F; Collaborative Study Group. Feasibility, safety, and short-term outcome of leadless ultrasound-based endocardial left ventricular resynchronization in heart failure patients: results of the wireless stimulation endocardially for CRT (WiSE-CRT) study. Europace. 2014 May;16(5):681-8. doi: 10.1093/europace/eut435. Epub 2014 Feb 4. PMID 24497573
- [Derived] Auricchio A, Delnoy PP, Regoli F, Seifert M, Markou T, Butter C; collaborative study group. First-in-man implantation of leadless ultrasound-based cardiac stimulation pacing system: novel endocardial left ventricular resynchronization therapy in heart failure patients. Europace. 2013 Aug;15(8):1191-7. doi: 10.1093/europace/eut124. Epub 2013 May 23. PMID 23703364